CLINICAL TRIAL: NCT03208816
Title: Community-Led Action Research in Oncology: Improving Symptom Management
Acronym: CLARO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Kathleen Lyons, PI, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CPHS30340
Record Dates: First submitted 2017-06-22; First posted 2017-07-06 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Chemotherapy-induced Neutropenia; Chemotherapy-induced Nausea and Vomiting; Anxiety; Depression; Fatigue; Neoplasms
Keywords: pain; constipation
MeSH Terms: conditions — Vomiting; Anxiety Disorders; Depression; Fatigue; Neoplasms; Pain; Constipation

STUDY DESIGN:
Intervention Model Description: a non-pharmacological, telephone-delivered, symptom management program for chemotherapy patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Other): symptom management program for chemotherapy patients
  Interventions: Behavioral: symptom management program for chemotherapy patients

INTERVENTIONS:
Behavioral: symptom management program for chemotherapy patients — Nurses will call study participants two times a week, to proactively assess and manage symptoms they might be experiencing during chemotherapy.

SUMMARY:
This study will be conducted at La Liga Contra el Cancer in San Pedro Sula, Honduras. The overall objective of this project is to improve symptom management for patients undergoing chemotherapy in Honduras. The first step in this line of research is a "proof of concept" feasibility study in which the investigators will demonstrate their ability to train nurses to administer a non-pharmacological, telephone-delivered, symptom management program for chemotherapy patients.

DETAILED DESCRIPTION:
The investigators will use the team's previous experience delivering a standardized, non-pharmacological palliative care intervention by telephone to inform a "proof of concept" feasibility study in Honduras. They will train nurses at La Liga Contra el Cancer in San Pedro Sula to conduct the telephone sessions and monitor their fidelity to treatment as they enroll a minimum They will then evaluate the feasibility, acceptability, and potential effectiveness of the program.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are over the age of 18 and are beginning a chemotherapy regimen to treat any solid or hematological cancer will be eligible for the study.

Exclusion Criteria:

* Patients who do not start planned chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Recruitment feasibility | Through study completion , an average of one year
  Number patients enrolled in the study divided by number of patients referred to the study

SECONDARY OUTCOMES:
Intervention feasibility | Through study completion, an average of one year
  Average number of minutes for each telephone sessions
Fidelity to treatment | Through study completion, an average of one year
  Average fidelity score for rated telephone sessions
Acceptability of intervention | At study completion, approximately one year
  Semi-structured interview of patients and nurse interventionists
Healthcare utilization | 12 weeks after enrollment
  Average number of cancelled appointments, emergency room visits, and toxicity requiring change in treatment plan

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen D Lyons, ScD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (2):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States
- La Liga Contra el Cancer, San Pedro Sula, Honduras

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bejarano S, Freed ME, Zeron D, Medina R, Zuniga-Moya JC, Kennedy L, Bruce ML, Zubkoff L, Bakitas MA, Lyons KD. Feasibility of a Symptom Management Intervention for Honduran Adults Undergoing Chemotherapy. West J Nurs Res. 2019 Oct;41(10):1517-1539. doi: 10.1177/0193945918825374. Epub 2019 Feb 12. PMID 30755109